CLINICAL TRIAL: NCT01508897
Title: A Randomized, Single-blind, Single-centre, Two-period, Cross-over Trial Investigating the Bioequivalence Between Completed Phase 2 and Planned Phase 3 Formulations of Liraglutide in Healthy Subjects
Brief Title: Comparison of Two Liraglutide Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NN2211-1331
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 2 formulation (Experimental)
  Interventions: Drug: liraglutide
- Phase 3 formulation (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Single dose administered as subcutaneous injection
  Arms: Phase 2 formulation
Drug: liraglutide — Single dose administered as subcutaneous injection
  Arms: Phase 3 formulation

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to test for bioequivalence of two formulations of liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments
* Body Mass Index (BMI) of 18-27 kg/m^2 incl.

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the study, as judged by the investigator
* Impaired renal function
* Uncontrolled treated/untreated hypertension
* Any clinically significant abnormal ECG
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunodeficiency virus) antibodies
* History of alcoholism or drug abuse during the last 12 months
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the Investigator
* Excessive consumption of a diet deviating from a normal diet as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2004-05-28 (Actual); Primary Completion 2004-06-30 (Actual); Study Completion 2004-06-30 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) (0-t)
Cmax, maximum concentration

SECONDARY OUTCOMES:
AUC (0-infinity)
tmax, time to maximum concentration
t½, terminal half-life
Terminal elimination rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neu-Ulm, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com